CLINICAL TRIAL: NCT02306070
Title: Improving Treatment and Liver Fibrosis Outcomes With Metformin in HCV-HIV Co-infected and HCV Mono-infected Patients With Insulin Resistance.
Brief Title: Improving Fibrosis Outcomes With Metformin
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient funding
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTNPT 019
Record Dates: First submitted 2014-11-02; First posted 2014-12-03 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2017-09

CONDITIONS: HIV Infection; Hepatitis C
MeSH Terms: conditions — HIV Infections; Hepatitis C | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin + lifestyle modification (Experimental): Metformin + lifestyle modification pre, during and post HCV antiviral therapy
  Interventions: Drug: Metformin
- No Metformin + Lifestyle modification (Placebo Comparator): No metformin + lifestyle modification pre, during and post HCV antiviral therapy.
  Interventions: Drug: No metformin treatment

INTERVENTIONS:
Drug: Metformin — metformin treatment + standard of care dietary and exercise advice
  Other Names: lifestyle modification
  Arms: Metformin + lifestyle modification
Drug: No metformin treatment — no metformin treatment + standard of care dietary and exercise advice
  Other Names: lifestyle modification
  Arms: No Metformin + Lifestyle modification

SUMMARY:
This study will evaluate the role of Metformin on liver fibrosis in HCV-HIV co-infected and HCV mono-infected patients with insulin resistance receiving DAA HCV treatment.

DETAILED DESCRIPTION:
HCV antiviral therapy has evolved rapidly in recent years and access to these medications has improved. While SVR is associated with improved liver outcomes, the rate of liver fibrosis regression with SVR is variable and predictors of regression are not well established. In addition, achieving SVR in patients with cirrhosis does not necessarily prevent decompensation or eliminate the risk of HCC. A better understanding of the role insulin resistance and impaired glucose metabolism have on these outcomes in HCV patients who achieve SVR are needed.

Identifying and targeting potentially modifiable risk factors such as IR may be of significant importance in preventing progression of and promoting regression of liver fibrosis, reducing mortality and improving outcomes for HCV-HIV co-infected and HCV-mono-infected patients.

This proposed pilot study will be the first to evaluate the role of Metformin on liver fibrosis in HCV-HIV co-infected and HCV mono-infected patients with IR receiving DAA HCV treatment.

If Metformin is effective in reducing liver fibrosis in this patient population, this will represent a well-tolerated, easy to administer, inexpensive therapy that will protect against negative HCV outcomes. This study will also be an opportunity to evaluate the impact of insulin resistance and hyperglycemia have on viral clearance HCV-infected patients treated with interferon-free regimens. In addition, the study will further explore the relationship between HCV, insulin resistance and AFP levels.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 79 years old inclusive
2. Provision of informed consent
3. Documented history of chronic HCV RNA infection
4. Intending to start on any 8-12 week IFN-free HCV antiviral therapy
5. If HIV-infected and not on HIV antiretroviral therapy, a CD4 count at least > 200
6. Insulin resistance as determined by a HOMA-IR of > 2.0 at screening
7. Evidence of fibrosis on FibroScan® > 8.0 kPa, OR liver biopsy score > 2 (Batts-Ludwig System) [55] (within 2 years)

Exclusion Criteria:

1. Pregnant, suspected to be pregnant, planning to become pregnant or breastfeeding
2. Chronic HBV infection
3. HbA1c > 8.0
4. Use of immune suppressing medications
5. Active malignancy
6. Current or any previous treatment with Metformin, other oral diabetes medications,insulin
7. Pre-existing diabetes (type 1, type 2 or gestational diabetes)
8. Clinical evidence of decompensated cirrhosis (ascites, esophageal varices, hepatic encephalopathy, hepatocellular carcinoma)
9. Presence of renal impairment or when renal function is not known, and also in patients with serum creatinine levels above upper limit of normal range. Renal disease or renal dysfunction (e.g., as suggested by serum creatinine levels >= 136 umol/L (males), >= 124 umol/L (females) or abnormal creatinine clearance (60 mL/min))
10. History of congestive heart failure requiring pharmacologic therapy
11. Wilson's disease
12. Alpha-1 antitrypsin
13. Hemochromatosis
14. Biliary Cirrhosis
15. Alcohol consumption > 50 g / day on average (see Appendix B for conversion to volume)
16. Participation in other clinical investigations during the study
17. History of lactic acidosis, irrespective of precipitating factors

Active illicit drug use and stable health illness will not be exclusionary assuming it is unlikely to compromise study adherence to protocol and study drug. In HIV-infected participants, HIV antiretroviral use and suppressed HIV viral load will not be required for participation.

HCV antiviral therapy will not be withheld for any participant that is eligible and desires to start treatment. If HCV treatment is anticipated to be started during the 48-week period of assessment, then participants will not be enrolled.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-09-30 (Actual); Study Completion 2018-04-03 (Estimated)

PRIMARY OUTCOMES:
Change in FibroScan® score (kPa) from baseline to week 12 (start of HCV treatment), compared between treatment groups. | 12 weeks
  liver elastography score (kPa)

SECONDARY OUTCOMES:
Virological response rates (SVR 12 weeks post HCV antiviral therapy) between treatment groups. | 12 weeks
  HCV RNA level (IU/mL)
Change in APRI measurements from baseline compared between treatment groups. | 12, 24, 48weeks
  calculated APRI
Change from baseline in glucose metabolism (HOMA-IR, fasting insulin, glucose levels) | 4, 8, 12, 24, 36, 48 weeks
  fasting glucose and insulin
Changes from baseline in lipid levels | 12, 36, 48 weeks
  fasting total cholesterol, LDL-c, HDL-c, triglycerides
Changes from baseline in anthropometric measures | 4, 8, 12, 24, 36, 48 weeks
  waist circumference, body weight and BMI
Changes from baseline in liver-related inflammatory markers | 4, 8, 12, 24, 36 weeks
  IL-6, IL-8, TNF-alpha, TGF-beta, C-reactive protein
Changes in AFP levels from baseline | 12, 24, 36, 48 weeks
  AFP
Participant acceptability to study medication dosing (in Arm 1 only) | 8, 24, 48 weeks
  Participant acceptability will be evaluated in Arm 1 only using the Treatment Satisfaction Questionnaire for Medication (TSQM), Version 1.4
Changes from baseline in diet | 24, 48 weeks
  Changes in diet from baseline will be captured using the International Physical Activity Questionnaire short-form (IPAQ-sf)
Changes from baseline in physical exercise parameters | 24, 48 weeks
  Changes in physical activity from baseline will be captured using the International Physical Activity Questionnaire short-form (IPAQ-sf)

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Cooper, MD, Principal Investigator — The Ottawa Hospital Division of Infectious Diseases
Locations (1):
- The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Doyle MA, Singer J, Lee T, Muir M, Cooper C. Improving treatment and liver fibrosis outcomes with metformin in HCV-HIV co-infected and HCV mono-infected patients with insulin resistance: study protocol for a randomized controlled trial. Trials. 2016 Jul 20;17(1):331. doi: 10.1186/s13063-016-1454-6. PMID 27439433
- See also: CIHR Canadian HIV Trials Network — http://www.hivnet.ubc.ca/home/